CLINICAL TRIAL: NCT02020304
Title: Effect of Temperature of Combined Spinal Epidural Dosing on Duration
Brief Title: Combined Spinal-Epidural Temperature and Duration of Action
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB 23933
Record Dates: First submitted 2013-11-21; First posted 2013-12-24 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Pain
Keywords: Combined spinal epidural duration; labor pain
MeSH Terms: conditions — Pain; Labor Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Room temperature (Experimental): room temperature combined spinal epidural dose (60-75 degrees F)
  Interventions: Drug: combined spinal epidural
- refrigerated temperature (Active Comparator): refrigerated temperature combined spinal epidural dose (~<43 degrees F)
  Interventions: Drug: combined spinal epidural

INTERVENTIONS:
Drug: combined spinal epidural — Combined Spinal Epidural

SUMMARY:
The hypothesis is that a combined spinal-epidural drug at refrigerated temperature will have a shorter period of pain relief than that maintained at room temperature. The temperature of the dose of medication will be measure with an infrared thermometer immediately prior (within 5 minutes) to administration.

DETAILED DESCRIPTION:
Subjects will receive a combined spinal epidural medication as per standard of care to treat their labor pain; however, they will be randomized to receive either a dose maintained at room temperature (60-75 degrees F) or one maintained in a refrigerator (~<43 degrees F). Duration of action will be done by assessments of pain, vital signs, nausea, itching, bromage and fetal heart rate every 15 minutes until the subject requests additional pain medication to treat their labor pain.

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years of age not allergic to medications used to treat labor pain </= 6cm cervical dilation visual pain score >/=3

Exclusion Criteria:

* <18 years of age > 6 cm cervical dilation non-English speaking subjects

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2013-08-29 (Actual); Primary Completion 2014-05-04 (Actual); Study Completion 2014-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vernon Ross, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Forsyth Medical Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Room Temperature | Refrigerated Temperature
Started | 30 | 28
Completed | 27 | 26
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Room Temperature | Refrigerated Temperature | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 26 | 53
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 53
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: Time
Description: length of time in minutes the combined spinal epidural dose duration is calculated from the time of administration until the request is made for additional analgesia (~1.5-3 hours) post dose. The subjects epidural is then dosed as per standard of care.
Time Frame: up to 3 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Room Temperature | Refrigerated Temperature
Number analyzed (Participants) | 27 | 26
minutes | 74 (29) | 81 (32)

2. Secondary Outcome: Analgesia Onset-5 Minutes Post Injection
Time Frame: from time of CSE administration
Population: number of subjects who achieved a VAS pain score of </=3 at 5 minutes after CSE injection
Measure: Count of Participants; unit: Participants
Arm/Group | Room Temperature | Refrigerated Temperature
Number analyzed (Participants) | 27 | 26
Participants | 24 | 14

3. Secondary Outcome: Analgesia Onset-10 Minutes Post Injection
Time Frame: up to 3 hours
Population: number of subjects who achieved a VAS pain score of </= 3 at 10 minutes after CSE injection
Measure: Count of Participants; unit: Participants
Arm/Group | Room Temperature | Refrigerated Temperature
Number analyzed (Participants) | 27 | 26
Participants | 25 | 19

4. Secondary Outcome: Analgesia Onset-15 Minutes Post Injection
Time Frame: up to 3 hours
Population: number of subjects who achieved a VAS pain score of </= 3 at 15 minutes after injection
Measure: Count of Participants; unit: Participants
Arm/Group | Room Temperature | Refrigerated Temperature
Number analyzed (Participants) | 27 | 26
Participants | 25 | 24

5. Secondary Outcome: Pruritus
Description: patients reporting pruritis at 30 minutes after CSE injection, self reported and measured on a scale of 0 (no itching at all) up to 10 (itching as bad as can be imagined)
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Room Temperature | Refrigerated Temperature
Number analyzed (Participants) | 27 | 26
units on a scale | 2 (1) | 1 (2)

ADVERSE EVENTS:
Time Frame: up to 3 hours after dosing
Arm/Group | Room Temperature | Refrigerated Temperature
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 0/27 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes